CLINICAL TRIAL: NCT06294613
Title: A Prospective, Open-label, Single-center, Study of the ACUSURGICAL Luca System for Treatment of Vitreoretinal Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acusurgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIV-23-07-043672
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-02

CONDITIONS: Vitreoretinal Disease
MeSH Terms: interventions — Vitreoretinal Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- vitreoretinal surgery supported by Luca System (Other)
  Interventions: Device: vitreoretinal surgery

INTERVENTIONS:
Device: vitreoretinal surgery — Patients undergoing vitreoretinal surgery

SUMMARY:
Prospective, interventional, open-label, non-controlled, monocentric study in Belgium of Luca, of up to 15 evaluable subjects, undergoing vitreoretinal surgery to treat intravitreal hemorrhage and macular pucker.

Only one eye per subject can be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Given written Informed Consent by subject,
* Males or females aged 18 - 85 years, pseudophakic or aphakic,
* Willing and able to comply with the schedule for follow-up visits,
* Requiring vitrectomy under general anesthesia (conditions include vitreous hemorrhage treatment (with potential clinical conditions including diabetic retinopathy, vascular occlusion, adverse effect of anticoagulant therapy), macular pucker),
* BCDVA <7/10,
* Deemed fit for robotic surgery per surgeons' assessment, including ability to undergone general anesthesia,
* Beneficiary of health insurance.

Exclusion Criteria:

* Uncontrolled systemic disease that could increase the operative risk or confound the outcome (autoimmune disease, uncontrolled hypertension, lung and heart disease impairing respiratory function, or any other medical condition as deemed by the Clinical Investigator),
* BMI (kg/m²) > 30,
* Axial length <22 or >26 mm per ocular biometry, inclusive,
* Presence of clinically significant ocular inflammation or infection within 30 days of Preop Visit, such as CME, uveitis, etc.,
* Ocular condition, that in the opinion of the Clinical Investigator, may predispose for future complications or confound visual acuity results, including profound amblyopia (<1/10) or strabismus,
* Ocular condition presenting associated pathology likely to require additional surgical manipulation, such as known need for membrane peeling, or retinal neovacular formation to be cut,
* Already vitrectomized on the study eye,
* Presenting retinal detachment or retinal tear,
* History of ocular traumatism; post-traumatic vitreous hemorrhage,
* Corneal scar preventing clear visualization of fundus,
* Any associated ocular pathology or ocular degenerative disorder that is uncontrolled such as glaucoma with clinical visual defect or IOP not controlled by medical treatment, uveitis, optic nerve damage,
* Subjects without light perception,
* Subject participating in other clinical studies,
* Subject being dependent on the Sponsor or Clinical Investigator,
* Pregnant or lactating women, based on self-declaration.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Safety Outcome | 3 Months
  incidence and severity of investigational device-related (definitely or probably) adverse events, for all subjects treated with the study device (Safety Population).

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Gent, Ghent, East Flanders, Belgium